CLINICAL TRIAL: NCT03481153
Title: Post-concussion and Transcranial Direct Current Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Naznin Virji-Babul, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBColumbia
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham tDCS (Placebo Comparator): Participants will be participate in a 20-minute sham tDCS session. tDCS electrodes will be placed on the left (anodal positive polarity) and right (cathodal;negative polarity) dorsolateral prefrontal cortex. Sham stimulation will be applied.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- tDCS (Active Comparator): Participants will participate in a 20-minute tDCS session. tDCS electrodes will be placed on the left (anodal positive polarity) and right (cathodal;negative polarity) dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — tDCS is a safe, non-invasive neurostimulation technique that can modulate neural excitability in the brain to positively impact cognition, behaviour and mood, particularly when combined with a behavioural intervention

SUMMARY:
Children and youth are at a greater risk of concussions than adults, and once injured, take longer to recover. The increased incidence of sports-related concussion in youth and the potentially serious long-term negative impact on their developing brains has enormous repercussions. While most young athletes recover within several days, many continue to experience symptoms for many months post-concussion. Symptoms are wide ranging and include - most notably: headache, sleep disturbances, brain fog, irritability as well as impairments in emotion and cognitive function (i.e. attention, memory, concentration, etc.). Yet there are no evidence-based intervention studies that have successfully addressed these symptoms. Thus, there is an urgent need for improved therapeutic strategies, which promote optimal functional recovery in youth concussion.

Transcranial direct current stimulation (tDCS) is a safe, non-invasive neurostimulation technique that can modulate neural excitability in the brain to positively impact cognition, behaviour and mood, particularly when combined with a behavioural intervention. Our long-term goal is to determine whether exercise combined with neurostimulation improves recovery from concussion. However, to our knowledge, the therapeutic potential of tDCS has not been studied in youth with concussion. Our objectives are as follows:

1. To determine the tolerability of a 20-minute session of tDCS in symptomatic youth athletes;
2. To evaluate the association between symptoms and EEG metrics at baseline and following a single session of tDCS in symptomatic athletes and compare these associations in symptomatic athletes who do not receive tDCS.

DETAILED DESCRIPTION:
Transcranial direct current stimulation is a non-invasive technique of neuromodulation that is inexpensive, easy to use and more importantly shows great promise to modify cortical excitability. Application of a weak direct current through the scalp has been shown to induce polarity specific changes in the excitability of cortical neurons23. This effect of transcranial direct current stimulation was first demonstrated in the human motor cortex. Since then it has also shown to be effective for other brain regions such as visual, somatosensory or frontal regions.

The advantage of tDCS in managing concussion is that this technique can be used to focally suppress or enhance neuronal firing depending on the size and location of the applied electrodes. Thus, at different points during the trajectory of concussion, the technique can be matched to the underlying pathophysiology. For example, work by Demitras et al suggests that cathodal tDCS may be used to suppress the acute glutamatergic hyperexcitability in the acute stages of brain injury; in the subacute stage, when GABAergic activity is excessive, anodal tDCS may increase excitability to counter these aberrant GABAergic effects. In the chronic stage, brain stimulation coupled to rehabilitation may enhance behavioral recovery, learning of new skills and cortical plasticity. Thus far, one pilot study has shown that a single session of anodal tDCS over the dorsolateral prefrontal cortex was associated with improvements in attention in adults with chronic TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic youth athletes (between18-25 years) who are between one to three months post concussion (participants will have had a witnessed head impact during a practice or game and be diagnosed with a concussion by team medical staff).
2. Regular participation in organized sport (>2 practice or games per week)

Exclusion Criteria:

1. No history of a developmental disorder.
2. No prior moderate-to-severe traumatic brain injury.
3. Fewer than four lifetime concussions (any cause),
4. No diagnosis or family history of schizophrenia, major depressive disorder, bipolar disorder or other psychiatric diagnosis
5. no previous history of seizures.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Comfort Rating Questionnaire (CRQ) | 10 minutes
  The scale asks participants to rate the following during and after the stimulation on a scale from 1-10 with 1 = not all all and 10= extremely: pain, tingling, burning, fatigue, nervousness, disturbed concentration, disturbed visual perception, headache. Three additional questions (yes/no response) are also asked: 1) Was the stimulation uncomfortable, 2)Did you notice a flash during/after the stimulation and 3) Did you notice sleep disturbances after the stimulation?

SECONDARY OUTCOMES:
Symptom checklist from the Sports Assessment Concussion Assessment Tool - 5th Edition | 10 minutes
  Participants are asked to indicate the symptom severity of 22 symptoms on the checklist. The scores range from 0 (none) to 6 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Naznin Virji-Babul, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided